CLINICAL TRIAL: NCT04893694
Title: the Prevalence of Oral Manifestation in Patients With SARS-CoV2 Infection
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Collaborators: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Other Study IDs: Oral SARS 2
Record Dates: First submitted 2021-05-15; First posted 2021-05-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV2; Oral Manifestation; prevalence
MeSH Terms: conditions — COVID-19; Oral Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-Cov2 virus was identified in china at the end of 2019 and spread worldwide causing a global pandemic. Current research showed that SARS-Cov2 virus invades human cells via the receptor angiotensin-converting enzyme 2 (ACE2) through scRNA-seq data analyses. The study identified the organs that are at risk and are vulnerable to SARS-CoV-2 infection. Therefore, cells with ACE2 receptor distribution may become host cells for the virus and cause inflammatory response in related organs and tissues, such as the tongue mucosa and salivary glands. These results suggest that oral mucosa could be a target of SARS-CoV-2 infection

DETAILED DESCRIPTION:
The oral cavity is particularly susceptible to viral infection with several viruses such as herpes simplex virus, cytomegalovirus and Zika virus because of its structures, especially salivary glands and soft tissues . Moreover, oral mucosa can be affected by secondary pathological process of a bacterial or fungal nature due to viral immunosuppression. The oral cavity could be considered a "biological barometer" of both viral infection and viral immunosuppression advancement .

The SARS-Cov2 virus was identified in china at the end of 2019 and spread worldwide causing a global pandemic. Current research showed that SARS-Cov2 virus invades human cells via the receptor angiotensin-converting enzyme 2 (ACE2) through scRNA-seq data analyses. The study identified the organs that are at risk and are vulnerable to SARS-CoV-2 infection. Therefore, cells with ACE2 receptor distribution may become host cells for the virus and cause inflammatory response in related organs and tissues, such as the tongue mucosa and salivary glands. These results suggest that oral mucosa could be a target of SARS-CoV-2 infection .

Although many authors reported the presence of oral lesion associated with SARS-CoV2 infection, the prevalence of the oral manifestation and the range of oral manifestation are still unknown. Further studies are necessary to better understanding of the symptoms of the SARS-CoV2 virus in order to faster detection. A multidisciplinary team following the patients could be the key in treatment of the infection and faster recovery.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of SARS-CoV2 with PCR.
* Age range from 18-60 years old
* Hospital admission not more than 10 days

Exclusion Criteria:

* Pregnancy or contraceptive pills
* Lactation
* Any auto-immune disease that could affect the oral mucosa
* On any neoplastic therapy.
* Uncontrolled diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is a multicenter cross- sectional study to study the prevalence of oral manifestation among patients with SARS-CoV2 infection and identify the range of the oral manifestation and site of lesions
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Oral Manifestation | one week
  presence or absence of Oral Manifestation in SARS-CO2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu H, Zhong L, Deng J, Peng J, Dan H, Zeng X, Li T, Chen Q. High expression of ACE2 receptor of 2019-nCoV on the epithelial cells of oral mucosa. Int J Oral Sci. 2020 Feb 24;12(1):8. doi: 10.1038/s41368-020-0074-x. PMID 32094336
- [Background] Dziedzic A, Wojtyczka R. The impact of coronavirus infectious disease 19 (COVID-19) on oral health. Oral Dis. 2021 Apr;27 Suppl 3(Suppl 3):703-706. doi: 10.1111/odi.13359. Epub 2020 May 6. PMID 32304276
- [Background] Riad A, Klugar M, Krsek M. COVID-19-Related Oral Manifestations: Early Disease Features? Oral Dis. 2022 Apr;28 Suppl 1(Suppl 1):940-942. doi: 10.1111/odi.13516. Epub 2020 Jul 16. No abstract available. PMID 32603497